CLINICAL TRIAL: NCT05973526
Title: Comparative Acute Effects of the Application of Percutaneous and Transcutaneous Electrolipolysis on the Female Abdominal Contour: a Cross Over Clinical Trial
Brief Title: Comparison of the Effects of Electric Current With Needles and Surface Electrodes on the Abdominal Contour of Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Principal Investigator, Rennatha de Moura Medeiros, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Eletrolipolysis
Record Dates: First submitted 2023-07-21; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Abdominal Fat
Keywords: adipose tissue; subcutaneous fat

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous (Experimental): In one of the infraumbilical hemibody, for percutaneous electrolipolysis, 2 pairs of needles will be introduced (0 ,25mm x 40mm) paired at a distance of 5 cm at 45º reaching the dermis-hypodermis tissue. The needles will be positioned at a distance of 2 cm laterally to the umbilicus and 5 cm below this marking, covering an area of about 10 cm laterally. This technique will have their electrodes connected to the Neurodyn 10-channel device belonging to the brand Ibramed®, in the electrolipolysis program.
  Interventions: Procedure: Percutaneous Electrolipolysis
- Transcutaneous (Experimental): In one of the infraumbilical hemibody, for transcutaneous electrolipolysis, 1 pair of silicone electrodes with conductive gel will be fixed with adhesive tape. The surface electrodes will be positioned at a distance of 2 cm laterally to the umbilicus and 5 cm below this marking, This technique will have their electrodes connected to the Neurodyn 10-channel device belonging to the brand Ibramed®, in the electrolipolysis program.
  Interventions: Procedure: Transcutaneous Electrolipolysis

INTERVENTIONS:
Procedure: Percutaneous Electrolipolysis — Electrolipolysis consists in the passage of electric current to the adipose tissue, causing lipolysis. The proposed protocol consists of 2 weekly sessions for 6 weeks, totaling 12 sessions, using needles.
  Arms: Percutaneous
Procedure: Transcutaneous Electrolipolysis — Electrolipolysis consists in the passage of electric current to the adipose tissue, causing lipolysis. The proposed protocol consists of 2 weekly sessions for 6 weeks, totaling 12 sessions, using the surface electrodos.
  Arms: Transcutaneous

SUMMARY:
The goal of this clinical trial is to compare the acute effects of percutaneous and transcutaneous eletroclipolysis on abdominal contour in women. The main question it aims to answer are:

• Is there superiority in percutaneous and transcutaneous electrolipolysis techniques?

Participants will undergo 12 sessions of 50 minutes each performed twice a week, totaling 6 weeks, after randomizing the hemibody for each technique.

Researchers will compare the hemibody with the percutaneous technique with the hemibody with the transcutaneous technique to see if there is a reduction of the adipose tissue.

DETAILED DESCRIPTION:
Abdominal Adiposity consists of an increase in adipose tissue in the abdomen region, which may be associated as a risk factor for cardiovascular pathologies, metabolic disorders and dyslipidemias, in addition to affecting self-esteem and social life due to aesthetics body provided by the volume increase of the contour. Electrolipolysis proves to be one of the accessible and low-cost resources, capable of promoting good therapeutic results through the passage of electric current to the adipose tissue, either with its percutaneous or transcutaneous technique. The study aims to compare the acute effects of percutaneous and transcutaneous electrolipolysis, considering comfort during execution.

ELIGIBILITY:
Inclusion Criteria:

* Women between with localized abdominal fat
* Body Mass Index (BMI) between 18.5 and 29.9 kg/m2 (adequate weight and overweight)
* Who have not undergone any treatment for the condition experienced in the last 6 months
* Sedentary
* Not on a supervised diet

Exclusion Criteria:

* Smokers
* Alcoholics
* Pregnant women
* Metabolic and circulatory system disorders
* Pacemaker
* Metallic implants
* Tumors/metastasis
* Dermatitis
* In treatment with corticosteroids and/or prolonged progesterone
* Skin ulcers/lesions
* Needle phobia (aichmophobia)
* Sensitivity alteration in the region to be treated
* Unable to understand the form and/or procedure
* Not completing the suggested protocol
* Dietary changes during the research

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of Adipose Tissue | From enrollment to end of treatment at 6 weeks
  It is expected to find a reduction in adipose tissue in both techniques, with similar results, verified by ultrasonography and adipometry, from the verification of a variation in the pre- and post-intervention measurements of thickness of adipose tissue in centimeters

SECONDARY OUTCOMES:
Vascularization Changes | From enrollment to end of treatment at 6 weeks
  Evaluate the possible alterations in the vascularization of the infraumbilical region through thermography, from the verification of variation in the pre- and post-intervention measures in body temperature in degrees celsius.
Satisfaction Evaluation | From enrollment to end of treatment at 6 weeks
  Evaluate satisfaction with each technique using a Likert-type scoring scale. The satisfaction scale ranges from 1 to 5, where 1 is the worst score and means no satisfaction, and 5 is the best score, extremely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Renato Guerino, PhD, Study Director — Physical Therapy Department, Universidade Federal de Pernambuco; Juliana Netto Maia, PhD, Study Director — Physical Therapy Department, Universidade Federal de Pernambuco
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Background] AROCA, Graciele Guimarães Pitelli et al. Thermographic and anthropometric assessment of electrical stimulation on localized body fat. Fisioterapia em movimento, v. 30, p. 29-37, 2017.
- [Background] CASTILLO, Carlos et al. Efeitos imediatos do ultrassom estacionário sobre a gordura subcutânea e retenção hídrica na região abdominal. Revista Inspirar Movimento & Saude, v. 22, n. 2, 2022.
- [Background] MELLO, Pâmela Billig et al. Comparação dos efeitos da eletrolipólise transcutânea e percutânea sobre a gordura localizada na região abdominal e de flancos através da perimetria e análise de bioimpedância elétrica. Fisioterapia Brasil, v. 11, n. 3, p. 198-203, 2010.
- [Background] CUNHA, Marisa; CUNHA, Ana Lucia; MACHADO, Carlos. Fisiopatologia da lipodistrofiaginoide. Surgical&Cosmetic Dermatology., v. 7, n. 2, p. 98-102 2015.
- [Background] EÇA, Lilian Piñeiro Marcolin et al. Estudo histológico comparativo e controlado de fibras colágenas da pele humana após terapia celular com fibroblastos. Surgical&Cosmetic Dermatology, v. 7, n. 3, p. 206-210, 2015.
- [Background] Feng B, Zhang T, Xu H. Human adipose dynamics and metabolic health. Ann N Y Acad Sci. 2013 Apr;1281(1):160-77. doi: 10.1111/nyas.12009. Epub 2013 Jan 14. PMID 23317303
- [Background] FERREIRA, Susan Caroline Santos et al. Ação e eficácia do tratamento com a Radiofrequência na adiposidade abdominal em mulheres. Revista de psicologia, v. 11, n. 38, p. 349-358, 2017.
- [Background] GONÇALVES, Michel Moraes et al. Alterações fisiológicas, percepção subjetiva de esforço e percepção de conforto durante formatura militar: um estudo experimental. Revista de Educação Física/Journal of Physical Education, v. 88, n. 3, 2019.
- [Background] Grabner GF, Xie H, Schweiger M, Zechner R. Lipolysis: cellular mechanisms for lipid mobilization from fat stores. Nat Metab. 2021 Nov;3(11):1445-1465. doi: 10.1038/s42255-021-00493-6. Epub 2021 Nov 19. PMID 34799702
- [Background] Guglielmi V, Sbraccia P. Obesity phenotypes: depot-differences in adipose tissue and their clinical implications. Eat Weight Disord. 2018 Feb;23(1):3-14. doi: 10.1007/s40519-017-0467-9. Epub 2017 Dec 11. PMID 29230714
- [Background] Guth F, Bitencourt S, Bedinot C, Sinigaglia G, Tassinary JAF. Immediate effect and safety of HIFU single treatment for male subcutaneous fat reduction. J Cosmet Dermatol. 2018 Jun;17(3):385-389. doi: 10.1111/jocd.12466. Epub 2017 Dec 4. PMID 29205814
- [Background] Lee MJ, Wu Y, Fried SK. Adipose tissue heterogeneity: implication of depot differences in adipose tissue for obesity complications. Mol Aspects Med. 2013 Feb;34(1):1-11. doi: 10.1016/j.mam.2012.10.001. Epub 2012 Oct 13. PMID 23068073
- [Background] RIBEIRO, Ricardo et al. A ultrassonografia enquanto método para caracterização do tecido adiposo abdominal. Saúde & Tecnologia, n. 22, p. 13-21, 2019.
- [Background] SILVA, Julianna; ARAÚJO, Maria; GUERINO, Marcelo. The use of a thermographic camera in aiding the diagnosis of cellulite appearance. O mundo da saúde, v. 46, p. 279-288, 2022.
- See also: Thermographic and anthropometric assessment of electrical stimulation on localized body fat. — https://www.scielo.br/j/fm/a/GDJy5fQFJFvjggZP8rPk7wm/abstract/?lang=en
- See also: Efeitos imediatos do ultrassom estacionário sobre a gordura subcutânea e retenção hídrica na região abdominal. — http://revistams.inspirar.com.br/wp-content/uploads/2022/08/pub_1004-2021.pdf
- See also: Comparação dos efeitos da eletrolipólise transcutânea e percutânea sobre a gordura localizada na região abdominal e de flancos através da perimetria e análise de bioimpedância elétrica. — https://pesquisa.bvsalud.org/portal/resource/pt/lil-789764
- See also: Fisiopatologia da lipodistrofiaginoide. — https://www.redalyc.org/pdf/2655/265541072002.pdf
- See also: Estudo histológico comparativo e controlado de fibras colágenas da pele humana após terapia celular com fibroblastos. — https://www.redalyc.org/pdf/2655/265542585002.pdf
- See also: Human adipose dynamics and metabolic health. — https://pubmed.ncbi.nlm.nih.gov/23317303/
- See also: Ação e eficácia do tratamento com a Radiofrequência na adiposidade abdominal em mulheres. — https://idonline.emnuvens.com.br/id/article/view/900
- See also: Alterações fisiológicas, percepção subjetiva de esforço e percepção de conforto durante formatura militar: um estudo experimental. — https://revistadeeducacaofisica.emnuvens.com.br/revista/article/view/819
- See also: Lipolysis: cellular mechanisms for lipid mobilization from fat stores. — https://www.nature.com/articles/s42255-021-00493-6
- See also: Obesity phenotypes: depot-differences in adipose tissue and their clinical implications. — https://pubmed.ncbi.nlm.nih.gov/29230714/
- See also: Immediate effect and safety of HIFU single treatment for male subcutaneous fat reduction. — https://pubmed.ncbi.nlm.nih.gov/29205814/
- See also: Adipose tissue heterogeneity: implication of depot differences in adipose tissue for obesity complications. — https://pubmed.ncbi.nlm.nih.gov/23068073/
- See also: A ultrassonografia enquanto método para caracterização do tecido adiposo abdominal. — https://journals.ipl.pt/stecnologia/article/view/532
- See also: The use of a thermographic camera in aiding the diagnosis of cellulite appearance. — https://revistamundodasaude.emnuvens.com.br/mundodasaude/article/view/1386